CLINICAL TRIAL: NCT00790153
Title: A Randomized, Open, Two-Way Cross-Over, Single-Centre, Phase I Study to Assess the Counter Regulatory Response During Hypoglycaemia in Healthy Male Volunteers After a Single Oral Dose of AZD1656 Suspension in Comparison With Insulin Infusion
Brief Title: To Evaluate the Hormonal Response to Low Blood Sugar After a Single Oral Dose of AZD1656 Suspension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Klas Malmberg, MD, PhD, Prof. Medical Science Director, Emerging Products, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1020C00012
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes, hormonal response
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin; AZD1656

ARMS (2):
- 1 (Active Comparator): AZD1656
  Interventions: Drug: AZD1656
- 2 (Active Comparator): Insulin
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Insulin infusion given during 3 hours at one occasion.
  Arms: 2
Drug: AZD1656 — Single dose oral suspension given at one occasion.
  Arms: 1

SUMMARY:
To evaluate the hormonal response to low blood sugar after a single oral dose of AZD1656 suspension.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers.
* Clinically normal physical findings (incl. Electrocardiogram (ECG)) and laboratory values as judged by the investigator.
* Have a body mass index (BMI) ≥19 and ≤30

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the investigator, within 2 weeks before the first administration of the investigational product
* Intake of any prescribed medicine and OTC drugs (including herbals, vitamins and minerals), except for occasional paracetamol or nasal spray for nasal congestion, within two weeks before the first administration of the investigational product.
* Daily use of nicotine containing substances.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2008-11; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic variables | Blood samples taken repeatedly up to 6 hours during study days

SECONDARY OUTCOMES:
Pharmacokinetic variables | Blood samples taken repeatedly during 24 hours on study day sessions
Safety Variables (AEs, BP, pulse, electrocardiogram (ECG), hypoglycaemic symptoms and laboratory variables) | Taken repeatedly during treatment periods

CONTACTS AND LOCATIONS:
Overall Officials: Klas Malmberg, MD, PhD, Prof, Study Director — AstraZeneca R&D Mölndal; Linda Morrow, MD, Principal Investigator — Profil Institute for Clinical Research, Inc.
Locations (1):
- Research Site, Chula Vista, California, United States